CLINICAL TRIAL: NCT06351774
Title: An Adaptive Physiotherapy Intervention Augmented With a Healthy Mind Training Program for People With Chronic Low Back Pain
Brief Title: Project AdaPT: An Adaptive Physiotherapy Intervention Augmented With a Healthy Mind Training Program for People With Chronic Low Back Pain
Acronym: AdaPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio University (Other)
Collaborators: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 21-F-45
Record Dates: First submitted 2024-04-02; First posted 2024-04-08 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Back Pain Lower Back Chronic; Disability Physical
MeSH Terms: interventions — Physical Therapy Modalities; Meditation

STUDY DESIGN:
Intervention Model Description: A 2 armed sequential, multiple-assignment randomized trial design
Who Masked: Investigator
Masking Description: The investigator was masked to the initial treatment assignment. The outcome assessor was not masked to treatment assignment and monitored treatment response at the mid-intervention in order to recommend continuation of current treatment or to augment treatment with the Healthy Mind Innovations training program for individuals who did not favorably respond to standalone PT.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PT (Experimental): Participants will receive physiotherapy per clinical practice guideline recommendations for 8 weeks (Phase 1). At week 10, participants will complete the Oswestry Disability Index (ODI) to determine their response to treatment. Individuals who report a favorable response to PT, defined by a threshold of improvement of at least 30% in their ODI, will continue with their PT for an additional 8 weeks. Individuals who do not favorably respond to PT will receive the Healthy Minds Innovation (HMI) app for an additional 8 weeks (Phase 2).
  Interventions: Behavioral: Physical therapy
- PT+HMI (Experimental): Participants will receive physiotherapy per clinical practice guideline recommendations for 8 weeks, in addition to the Healthy Minds Innovation app (Phase 1). At week 10, participants will complete the Oswestry Disability Index (ODI) to determine their response to treatment. Individuals who report a favorable response to PT+HMI, defined by a threshold of improvement of at least 30% in their ODI, will continue with their PT+HMI for an additional 8 weeks. Individuals who do not favorably respond to PT+HMI will receive an in-person teacher-guided tai chi session and tai chi videos for guided self-practice for an additional 8 weeks (Phase 2).
  Interventions: Behavioral: Physical therapy

INTERVENTIONS:
Behavioral: Physical therapy — Physical therapy for the treatment of chronic low back pain, as directed by a licensed Physical Therapist. The Healthy Minds Innovations (HMI) program is an app-based learning platform developed through the University of Wisconsin-Madison Center for Healthy Minds. The HMI app includes foundational meditation practices and short podcast-style lessons based on the science of wellbeing to cultivate mindfulness, positive relationships, and insight into the nature of the self.
  Other Names: Meditation

SUMMARY:
In the proposed research, we will elucidate the comparative effectiveness of standalone physiotherapy (PT) vs. PT augmented with a self-guided, app-based Healthy Minds Innovation wellbeing program (PT+HMI) aimed at cultivating awareness, connection, insight, and purpose for people with chronic low back pain (CLBP).

DETAILED DESCRIPTION:
The overall objective is to primarily elucidate differential changes in CLBP patients administered PT or PT+HMI across physical health domains (back disability, pain interference, actigraphy, gait performance). Secondarily, we will elucidate changes in patient-reported physical health outcomes for early non-responders who go on to receive an adaptive intervention that provides augmented treatment pathways.

Our central hypothesis is that improvements in disability (primary outcome), i.e., responders to PT and PT+Well will be differentially associated with changes in physical activity levels, gait kinematics, psychological flexibility, and fear-avoidance. We further predict that initial non-responders who progress to augmented care will show improvements in the primary outcomes. We will conduct a two-armed RCT with 20 CLBP participants who will receive PT or PT+HMI and test our hypotheses in 3 specific aims. In Aim 1, we will use patient-reported measures of disability and pain interference to elucidate subjective physical health outcomes. In Aim 2, we will use actigraphy to measure physical activity levels, 3D trunk kinematic measures during gait, and a lifting task to reveal movement-based responders. In Aim 3, we will use patient-reported measures for indices of psychological flexibility and healthy emotionality to elucidate mental health processes that correlate with physical health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* A minimum age of at least 18 years; the ability to read and speak English; have visited a health care professional for back pain during the past 90 days with a physician referral for PT; have experienced back pain for at least 3 months duration and for at least ½ days in the past 6 months; and currently experiencing at least moderate back-related disability, which was operationalized as a score of ≥24% (12 out of 50 points) on the Oswestry Disability Index (ODI). Participants needed to have smart device access to engage with the HMI app.

Exclusion Criteria:

* Having undergone lumbar surgery within the past year; an ongoing disability or worker's compensation, or legal claim; informed by their physician the presence of a serious pathology causing their LBP; pregnancy or planning to become pregnant; and having previously received PT for LBP during the prior 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-05-24 (Actual); Primary Completion 2024-02-08 (Actual); Study Completion 2024-03-25 (Actual)

PRIMARY OUTCOMES:
Oswestry Disability Index | Baseline (T0), mid-treatment/week 10 (T1), post-treatment/week 26 (T2), and post-treatment/week 52 (T3)
  A self-reported outcome measure of back disability
PROMIS Pain Interference | Baseline (T0), post-treatment/week 26 (T2), and post-treatment/week 52 (T3)
  A self-reported outcome measure of pain interference

SECONDARY OUTCOMES:
Actigraphy | Baseline (T0) and post-treatment/week 26 (T2)
  Measure of physical activity levels for 10 days of home use
3D Motion Capture | Baseline (T0) and post-treatment/week 26 (T2)
  Trunk motion capture during walking and lifting tasks
Pain acceptance | Baseline (T0) and post-treatment/week 26 (T2)
  Chronic Pain Acceptance Questionnaire (CPAQ-20)
Committed action | Baseline (T0) and post-treatment/week 26 (T2)
  Committed Action Questionnaire (CAQ-8)
Healthy emotionality | Baseline (T0) and post-treatment/week 26 (T2)
  Emotional Styles Questionnaire (ESQ)
Exercise behavior | Baseline (T0), mid-treatment/week 10 (T1), post-treatment/week 26 (T2), and post-treatment/week 52 (T3)
  Stanford Exercise Behavior Scale (SEBS)
Back pain screening tool 1 | Baseline (T0)
  Örebro Musculoskeletal Pain Screening Questionnaire (ÖMPSQ-10)
Back pain screening tool 1 | Baseline (T0)
  Start Back Screening Tool (SBST-9)
Kinesiophobia | Baseline (T0)
  Tampa Scale of Kinesiophobia (TSK-11)
Attitudes towards complementary and alternative medicine | Baseline (T0)
  Healthcare Experiences and Attitudes List - Attitudes Towards Complementary and Alternative Medicine (HEAL-CAM)
Treatment expectancy | Baseline (T0)
  HEAL Treatment Expectancy (HEAL-TEX)
Lumbar pressure pain threshold | Baseline (T0) and week 26 (T2)
  Quantitative Sensory Testing
Thermal method of limits | Baseline (T0) and week 26 (T2)
  Quantitative Sensory Testing

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas V Karayannis, MPT, PhD, Principal Investigator — Ohio University
Locations (1):
- Ohio University, Athens, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided